CLINICAL TRIAL: NCT02312531
Title: HBIG for Prevention of Mother-to-infant HBV Transmission
Brief Title: Prevention for Mother-to-infant Transmission of HBV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, liu jinfeng, Xi'an Jiaotong University College of Medicine, Xi'an Jiaotong University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012ZX10002007-001-001 -1
Record Dates: First submitted 2014-12-02; First posted 2014-12-09 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: HBV
Keywords: HBV; Intrauterine infection; hepatitis B immunoglobulin; immune barrier; virus replication; placenta
MeSH Terms: interventions — hepatitis B hyperimmune globulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HBIG group (Experimental): Mothers in HBIG group received 'Hepatitis B immunoglobulin' (HBIG 200 IU, S20023028, Hualan Biological Engineering Inc.) injection at gestational weeks 20, 24, 28, 32, 34, 36, 38, 39, and 40.
  Interventions: Drug: Hepatitis B immunoglobulin
- Control group (No Intervention): Mothers in control group had no HBIG injection during pregnancy.

INTERVENTIONS:
Drug: Hepatitis B immunoglobulin — Hepatitis B immunoglobulin 200 IU injection at gestational week 20, 24, 28, 32, 34, 36, 38, 39, and 40 in HBIG group mothers.
  Other Names: HBIG
  Arms: HBIG group

SUMMARY:
In this study, HBV-infected pregnant women were divided into two groups, those who received and those who did not receive hepatitis B immunoglobulin (HBIG) during pregnancy. In the mothers, the changes in HBV serum markers (hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (HBsAb), HBeAg, hepatitis B core antibody (HBcAb)), and the DNA load were investigated. Immunohistochemical staining with custom-made antibodies against HBIG revealed both the level and distribution of HBIG in placentas. The protective mechanism of HBIG administrated during pregnancy was explored.

DETAILED DESCRIPTION:
Twenty-eight HBsAg-positive pregnant women who underwent consultation were recruited from the First Affiliated Hospital of Xi'an Jiaotong University, Shaanxi, China. Twelve of these women willing to receive HBIG administration were assigned to experimental group, while another sixteen without HBIG injection were enrolled as control group. The exclusion criteria for participants were: 1) infection with toxoplasmosis, syphilis, parvovirus B19, rubella, cytomegalovirus, herpes, hepatitis C, HIV, or other viruses; 2) obstetric diseases such as pregnancy-related hypertension, placental abruption, threatened miscarriage, and others.

The 12 pregnant women enrolled willing to receive injections of HBIG (200 IU, S20023028, Hualan Biological Engineering Inc.) beginning at week 20 of gestation (at weeks 20, 24, 28, 32, 34, 36, 38, 39, and 40). The control group only underwent regular examinations without any HBIG treatment during pregnancy. All the infants born received combined immunoprophylaxis (HBIG, 200 IU, and the first dose of the hepatitis B vaccine, 5 μg, S19983018, Shenzhen Kangtai Biological Products Co. Ltd.) at different injection sites within 12 h postpartum.

Data of mothers were collected from medical records that included complete healthcare information before and after delivery. Each infant was consecutively followed up after birth, growth index (weight, length and head circumference), feeding patterns and serum level of HBV DNA and viral markers were recorded. Serum HBV markers (HBsAg, HBsAb, HBeAg, and HBcAb) titers、HBV DNA load and liver function of mothers were regularly measured during pregnancy. Serum HBsAg, HBsAb titer and HBV DNA load of infants were tested at birth, the age of 7 and 12 months. Placental tissue sections were used for immunohistochemical staining of HBsAg (mouse, 1:50, ZM-0122, Beijing Zhongshan Golden Bridge Biotechnology Co.), HBIG (rabbit, 4.7 mg/ml, 1:2500, prepared as described above), and CD68 (mouse, 1:25, ab955, Abcam).

Adverse outcome, HBV infection rate of infants, HBV markers titers, liver function and HBV DNA load of mothers, correlation between mothers and newborns regarding HBsAb titer and histopathological changes in placenta samples were compared between experimental group and control group.

Statistical analysis was performed using SPSS 13.0 statistical software (SPSS Inc., Chicago, USA). Data were expressed as the mean ± standard deviation (SD). The data were analyzed with the Shapiro-Wilk test and the Levene statistic for normality and homogeneity of variance, respectively. The difference between two quantitative groups was compared with an independent-sample t-test or the Mann-Whitney U-test as appropriate, and correlations were analyzed with the Pearson or Spearman correlation test. The chi-square test or Fisher's exact test was used to compare the proportions of the two groups. All tests were two-tailed with the risk set at 5%, and the statistical significance was set as p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg positive for more than 6 months, gestational age less than 20 weeks

Exclusion Criteria:

* infection with toxoplasmosis, syphilis, parvovirus B19, rubella, cytomegalovirus, herpes, hepatitis C, HIV, or other viruses; obstetric diseases such as pregnancy-related hypertension, placental abruption, threatened miscarriage, and others.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
HBV infection of infants | one year
  HBV DNA and HBsAg positive at the age of 1 year old
Histopathological changes in placenta | at delivery
  Immunohistochemical staining of HBsAg, HBIG and CD68

SECONDARY OUTCOMES:
Serum HBV markers titers、HBV DNA load and liver function changes | at weeks 20, 24, 28, 32, 34, 36, 38, 39, and 40 of gestation
  Serum HBV markers (HBsAg, HBsAb, HBeAg, and HBcAb) titers、HBV DNA load and liver function of mothers were regularly measured.
Adverse events | at weeks 20, 24, 28, 32, 34, 36, 38, 39, and 40 of gestation, at delivery, at the age of 7 and 12 months of infants
  Reports of premature and partum complications, ALT flare, delivery mode and birth defects.

CONTACTS AND LOCATIONS:
Overall Officials: Tianyan Chen, MD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University